CLINICAL TRIAL: NCT03725228
Title: Lidocaine Compared to Magnesium Sulfate to Prolong Spinal Anesthesia: Non-inferiority Randomized Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Head of Anesthesia, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: tccRenato2018
Record Dates: First submitted 2018-10-27; First posted 2018-10-30 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Anesthesia; Pain
MeSH Terms: conditions — Pain | interventions — Magnesium Sulfate; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium Sulfate (Active Comparator): Continuous intravenous infusion of 15mg/kg/h of magnesium sulfate, starting just after spinal anesthesia infusion until the end of surgery
  Interventions: Drug: Magnesium Sulfate
- Lidocaine (Experimental): Continuous intravenous infusion of 1.5mg/kg/h of lidocaine, starting just after spinal anesthesia infusion until the end of surgery
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Magnesium Sulfate — Magnesium Sulfate 15mg/kg/h
  Arms: Magnesium Sulfate
Drug: Lidocaine — Lidocaine 1,5mg/kg/h
  Arms: Lidocaine

SUMMARY:
This study evaluates the addition of continuous infusion of lidocaine or continuous infusion of magnesium sufate in the duration of spinal anesthesia.

DETAILED DESCRIPTION:
Both lidocaine and magnesium sulfate have been shown to prolong spinal anesthesia.

The number of studies using magnesium sulfate to improve spinal anesthesia is greater than the number of studies using lidocaine, and methodology varies significantly between studies.

Adverse effects of lidocaine are different from magnesium sulfate's. Lidocaine has a wider therapeutic interval with fewer side effects, including: Drowsiness, Feeling Anxious, Feeling Cold, Nervous, Numbness And Tingling, Signs And Symptoms At Injection Site, Twitching.

Magnesium sulfate's side effects include: heart disturbances, breathing difficulties, poor reflexes, confusion, weakness, flushing (warmth, redness, or tingly feeling), sweating, lowered blood pressure, feeling like you might pass out, anxiety, cold feeling, extreme drowsiness, muscle tightness or contraction, or headache.

ELIGIBILITY:
Inclusion Criteria:

* Will receive spinal anesthesia for TURP por Histerectomy

Exclusion Criteria:

* Protocol violation;
* Severe adverse events;
* Change to general anesthesia or addition of epidural anesthesia;
* Complete or partial spinal block failure;
* Mental status alteration (agitation, confusion, loss of conciousness).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Sensitive block duration | 9 hours
  Thermal and pinprick level lowering to S2

SECONDARY OUTCOMES:
Motor block duration | 9 hours
  Time to Bromage return to baseline
Two levels regression | 9 hours
  Time from maximal thermal (cold) sensitive block level to lower two levels
Pain at postanesthesia care unit | 1-3 hours
  Maximum pain (0-10 verbal scale) during PACU

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário de Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified IPD in Mendeley Data after study completion
Supporting Information: Analytic Code
Time Frame: Analystic code will be published in RPUBS
Access Criteria: Open Access